CLINICAL TRIAL: NCT05964374
Title: Goal-Directed Therapy (GDT) Using Hypotension Prediction Index (HPI) Following Cardiac Surgery: a Pilot Randomized Control Trial
Brief Title: Goal-Directed Therapy Following Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB23-0043
Record Dates: First submitted 2023-06-21; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Surgery
Keywords: cardiac surgery; hemodynamic optimization; goal-directed therapy
MeSH Terms: interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Routine post-operative clinical care.
- Intervention (Experimental): Goal-directed therapy algorithm in addition to routine post-operative clinical care.
  Interventions: Device: Goal-directed therapy

INTERVENTIONS:
Device: Goal-directed therapy — Goal-directed therapy using HemoSphere® monitor, Acumen® transducer, and Hypotension Prediction Index® algorithm (Edwards Lifesciences, Irvine, USA),
  Arms: Intervention

SUMMARY:
Pilot prospective randomized control trial comparing goal-directed therapy algorithm vs routine care in the intensive care unit following cardiac surgery.

DETAILED DESCRIPTION:
Rationale:

Goal-directed therapy (GDT) has been shown to reduce complications and length of stay on cardiac surgery patients. Unfortunately, the existing literature on GDT in CV surgery has several limitations, which creates uncertainty over the expected benefit of implementing this care element with high associated costs and impact on workflow. Hypotension Prediction Index (HPI) is a proprietary algorithm that utilizes pulse contour analysis from invasive arterial pressure monitoring to identify patients at risk for becoming hypotensive within 15 minutes. The algorithm was developed using machine learning on a large surgical/ICU data set, and then externally validated on non-cardiac and cardiac surgical patients. HPI, as part of a GDT algorithm, may allow healthcare providers to identify patients recovering from cardiac surgery who may benefit from optimization prior to becoming hypotensive and assist with selecting the most appropriate hemodynamic intervention.

Hypothesis:

Application of an HPI-based GDT algorithm will result in a difference in cumulative fluid administration over the first 24-hours of index ICU admission following cardiac surgery.

Study Design:

Unblinded randomized controlled trial pilot. Data will be used to inform/justify the feasibility, design, and implementation of a future multi-center randomized controlled trial.

Study Population:

Moderate or high-risk (EuroSCORE II > 2%), non-emergent, adult open-heart cardiac surgery patients. Heart transplant, durable VAD implantation, or patients who require post-operative MCS support will be excluded.

Sample size= 100 (50 control : 50 intervention)

Intervention:

Patients randomized to the intervention arm will be monitored using the HPI technology and be treated following a GDT algorithm when HPI is >50 for 48-hours or duration of invasive arterial monitoring (whichever occurs first). The GDT algorithm is a standardized approach to identifying abnormal hemodynamic parameters and administering a prescribed therapy in a step-wise fashion with fixed re-assessment intervals (see attached).

What will be different from routine care? :

1. Hemodynamic interventions (fluid, inotropic, or vasopressor therapy) will be administered when HPI > 50 rather than MAP < 65.
2. Choice of applied therapy (fluid, inotropic, or vasopressor therapy) will be guided by a GDT algorithm.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Planned cardiac surgery using cardiopulmonary bypass (sternotomy or MICS)
3. Preoperative European System for Cardiac Operative Risk Evaluation II (EuroSCORE II) of 2% or more.
4. Informed consent obtained.

Exclusion Criteria:

1. Patients who refuse participation
2. Patients who are unable to give informed consent
3. Patients who are having a heart transplant or having surgery solely for an insertion of a ventricular assist device
4. Emergency surgery
5. Patients who require MCS (including ECMO, Impella, or IABP) post-operatively

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
24-hour cumulative IV fluid administration | 24-hours
  Cumulative post-operative intravenous fluid administration over the first 24-hours of index ICU admission.

SECONDARY OUTCOMES:
Fluid Administration | Duration of ICU stay, up to 30-days
  Daily average
Fluid Administration | Duration of ICU stay, up to 30-days
  Cumulative
Vasoactive medication administration | Duration of ICU stay, up to 30-days
  Daily average
Vasoactive medication administration | Duration of ICU stay, up to 30-days
  Daily cumulative
Vasoactive medication administration | Duration of ICU stay, up to 30-days
  Duration
Hemodynamic parameters | 48-hours or when arterial line removed
  Incidence of HPI > 50 greater than 5-minutes
Hemodynamic parameters | 48-hours or when arterial line removed
  Incidence of HPI > 85 greater than 5-minutes
Hemodynamic parameters | 48-hours or when arterial line removed
  Incidence of MAP < 65 greater than 5-minutes
Hemodynamic parameters | 24-hours
  Total Area Under the Curve (AUC) for HPI > 50
Hemodynamic parameters | 48-hours or when arterial line removed
  Total Area Under the Curve (AUC) for HPI > 50
Hemodynamic parameters | 24-hours
  Total Area Under the Curve (AUC) for HPI > 85
Hemodynamic parameters | 48-hours or when arterial line removed
  Total Area Under the Curve (AUC) for HPI > 85
Hemodynamic parameters | 24-hours
  Total Area Under the Curve (AUC) for MAP < 65
Hemodynamic parameters | 48-hours or when arterial line removed
  Total Area Under the Curve (AUC) for MAP < 65
Enrollment | 1-year
  Proportion of screened patients eligible for enrollment.
Enrollment | 1-year
  Proportion of eligible patients who consent to participate.
Study Protocol Compliance | 1-year
  Proportion of consented patients who complete all study assessments.
Arterial Monitoring Reliability | 1-year
  Number of arterial catheters requiring replacement
GDT algorithm compliance | 48-hours or when arterial line removed
  Time from HPI > 50 to application of an intervention
GDT algorithm compliance | 48-hours or when arterial line removed
  Proportion of hemodynamic interventions applied for HPI > 50 that were recommended by the algorithm
GDT algorithm compliance | 48-hours or when arterial line removed
  Proportion of hemodynamic interventions applied for MAP < 65 that would be recommended by the algorithm based on hemodynamic parameters.
GDT algorithm compliance | 48-hours or when arterial line removed
  MD notifications prompted by the GDT algorithm and resulting actions
GDT algorithm compliance | 48-hours or when arterial line removed
  Actions (therapies or investigations) prompted by an MD notification.
GDT algorithm compliance | 48-hours or when arterial line removed
  Number of study protocol suspensions
GDT algorithm compliance | 48-hours or when arterial line removed
  Duration of protocol suspensions
GDT algorithm compliance | 48-hours or when arterial line removed
  Rationale for protocol suspensions
End-organ dysfunction/injury | Index admission, up to 30-days
  Acute kidney injury
End-organ dysfunction/injury | Index admission, up to 30-days
  Delirium
End-organ dysfunction/injury | Index admission, up to 30-days
  Stroke
End-organ dysfunction/injury | Index admission, up to 30-days
  Ileus
End-organ dysfunction/injury | Index admission, up to 30-days
  Gut infarction
End-organ dysfunction/injury | Index admission, up to 30-days
  Prolonged mechanical ventilation (> 24 hours)
End-organ dysfunction/injury | Index admission, up to 30-days
  Deep sternal wound infection
End-organ dysfunction/injury | Index admission, up to 30-days
  Any surgical site infection
Transfusion | Index admission, up to 30-days
  Total red-blood cell administration
Transfusion | Index admission, up to 30-days
  Total fresh-frozen plasma administration
Transfusion | Index admission, up to 30-days
  Total platelet administration
Transfusion | Index admission, up to 30-days
  Total albumin administration
Mobilzation | Index admission, up to 30-days
  Time to first mobilization (dangle)
Mobilzation | Index admission, up to 30-days
  Time to first mobilization (stand)
Mobilization | Index admission, up to 30-days
  Time to first mobilization (walk)
Hydration | Index admission, up to 30-days
  Time to first PO hydration
Nutrition | Index admission, up to 30-days
  Time to first PO nutrition
Patient-centered Outcome | Index admission, up to 10-days
  Quality of Recovery-15 (QOR-15) at post-op days 3, 5, 7, and 10.
Patient-centered Outcome | Up to 1-year post-operative
  World Health Organization Disability Assessment Schedule (WHODAS 2.0) at baseline, 2-weeks, 30-days, 90-days, and 1-year.
Patient-centered Outcome | Up to 1-year post-operative
  MacNew Questionnaire at baseline, 2-weeks, 30-days, 90-days, and 1-year.
Patient-centered Outcome | Up to 1-year post-operative
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) at baseline, 2-weeks, 30-days, 90-days, and 1-year.
Patient-centered Outcome | 30-days
  Canadian Patient Experiences Survey on Inpatient Care (CPES-IC) at 30-days
Length of Stay | Up to 1-year post-operative
  ICU length of stay
Length of Stay | Up to 1-year post-operative
  Hospital length of stay
Re-admission | 30-days
  Incidence of hospital re-admission within 30-days of index surgery
Mortality | Up to 1-year post-operative
  7-day, 30-day, and 1-year mortality.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li P, Qu LP, Qi D, Shen B, Wang YM, Xu JR, Jiang WH, Zhang H, Ding XQ, Teng J. Significance of perioperative goal-directed hemodynamic approach in preventing postoperative complications in patients after cardiac surgery: a meta-analysis and systematic review. Ann Med. 2017 Jun;49(4):343-351. doi: 10.1080/07853890.2016.1271956. Epub 2017 Feb 2. PMID 27936959
- [Background] Osawa EA, Rhodes A, Landoni G, Galas FR, Fukushima JT, Park CH, Almeida JP, Nakamura RE, Strabelli TM, Pileggi B, Leme AC, Fominskiy E, Sakr Y, Lima M, Franco RA, Chan RP, Piccioni MA, Mendes P, Menezes SR, Bruno T, Gaiotto FA, Lisboa LA, Dallan LA, Hueb AC, Pomerantzeff PM, Kalil Filho R, Jatene FB, Auler Junior JO, Hajjar LA. Effect of Perioperative Goal-Directed Hemodynamic Resuscitation Therapy on Outcomes Following Cardiac Surgery: A Randomized Clinical Trial and Systematic Review. Crit Care Med. 2016 Apr;44(4):724-33. doi: 10.1097/CCM.0000000000001479. PMID 26646462
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Background] Hatib F, Jian Z, Buddi S, Lee C, Settels J, Sibert K, Rinehart J, Cannesson M. Machine-learning Algorithm to Predict Hypotension Based on High-fidelity Arterial Pressure Waveform Analysis. Anesthesiology. 2018 Oct;129(4):663-674. doi: 10.1097/ALN.0000000000002300. PMID 29894315
- [Background] Davies SJ, Vistisen ST, Jian Z, Hatib F, Scheeren TWL. Ability of an Arterial Waveform Analysis-Derived Hypotension Prediction Index to Predict Future Hypotensive Events in Surgical Patients. Anesth Analg. 2020 Feb;130(2):352-359. doi: 10.1213/ANE.0000000000004121. PMID 30896602
- [Background] Shin B, Maler SA, Reddy K, Fleming NW. Use of the Hypotension Prediction Index During Cardiac Surgery. J Cardiothorac Vasc Anesth. 2021 Jun;35(6):1769-1775. doi: 10.1053/j.jvca.2020.12.025. Epub 2020 Dec 21. PMID 33446404
- [Background] Parsons H, Zilahi G. Pro: Hypotension Prediction Index-A New Tool to Predict Hypotension in Cardiac Surgery? J Cardiothorac Vasc Anesth. 2023 Oct;37(10):2133-2136. doi: 10.1053/j.jvca.2023.05.023. Epub 2023 May 17. No abstract available. PMID 37301700
- [Background] Rellum SR, Schuurmans J, Schenk J, van der Ster BJP, van der Ven WH, Geerts BF, Hollmann MW, Cherpanath TGV, Lagrand WK, Wynandts P, Paulus F, Driessen AHG, Terwindt LE, Eberl S, Hermanns H, Veelo DP, Vlaar APJ. Effect of the machine learning-derived Hypotension Prediction Index (HPI) combined with diagnostic guidance versus standard care on depth and duration of intraoperative and postoperative hypotension in elective cardiac surgery patients: HYPE-2 - study protocol of a randomised clinical trial. BMJ Open. 2023 May 2;13(5):e061832. doi: 10.1136/bmjopen-2022-061832. PMID 37130670
- [Background] Maheshwari K, Buddi S, Jian Z, Settels J, Shimada T, Cohen B, Sessler DI, Hatib F. Performance of the Hypotension Prediction Index with non-invasive arterial pressure waveforms in non-cardiac surgical patients. J Clin Monit Comput. 2021 Feb;35(1):71-78. doi: 10.1007/s10877-020-00463-5. Epub 2020 Jan 27. PMID 31989416
- [Background] Baumgarten M, Brodsgaard A, Bunkenborg G, Foss NB, Norholm V. Nurse and Physician Perceptions of Working With Goal-Directed Therapy in the Perioperative Period. J Perianesth Nurs. 2020 Apr;35(2):198-205. doi: 10.1016/j.jopan.2019.09.005. Epub 2019 Dec 13. PMID 31843240